CLINICAL TRIAL: NCT06062329
Title: Evaluation of the Safety and Efficacy of the Symphony Thrombectomy System in the Treatment of Pulmonary Embolism
Brief Title: SYMPHONY-PE Study for Treatment of Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperative Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRU-2023-001
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Acute Pulmonary Embolism; Thromboembolism; Emboli, Pulmonary; Thrombosis; Thrombus; Embolism; Embolism; Cardiovascular Diseases; Vascular Diseases
Keywords: Thrombectomy; Submassive Pulmonary Embolism; Right Ventricle dysfunction
MeSH Terms: conditions — Thromboembolism; Pulmonary Embolism; Thrombosis; Embolism; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Symphony Thrombectomy system (Experimental): Mechanical thrombectomy using the Symphony Thrombectomy system for the treatment of acute pulmonary embolism.
  Interventions: Device: Symphony Thrombectomy System

INTERVENTIONS:
Device: Symphony Thrombectomy System — The Symphony Thrombectomy System will be used to restore blood flow to the pulmonary arteries by removing thrombus/embolus/clot using aspiration and mechanical clot engagement.

SUMMARY:
Evaluation of the Safety and Efficacy of the Symphony Thrombectomy System in the Treatment of Pulmonary Embolism

DETAILED DESCRIPTION:
SYMPHONY-PE is a pivotal study intended to assess the safety and efficacy of the Symphony Thrombectomy System to treat subjects with acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

1. CTA evidence of acute PE within ≤14 days
2. Clinical signs and symptoms consistent with acute PE.
3. Systolic BP ≥90 mmHg with evidence of dilated RV with an RV/LV ratio >0.9 (based on Investigator's assessment of RV/LV ratio)
4. Stable heart rate <130 BPM prior to procedure
5. Subject is between 18 and 80 years of age
6. Subject is willing to sign an IRB-approved informed consent form
7. Subject is willing and able to comply with protocol follow-up

Exclusion Criteria:

1. Thrombolytic use within 14 days of baseline CTA
2. International Normalized Ratio (INR) >3
3. Platelets <100,000/µL
4. Kidney dysfunction as confirmed by serum creatinine >1.8 mg/dL or GFR <45 mL/min
5. Hematocrit <28% or hemoglobin <9 g/dL
6. Systolic BP <90 mmHg for 15 min or requirement of inotropic support to maintain systolic BP ≥90 mmHg any time after admission
7. Experienced cardiac arrest
8. Has left bundle branch block
9. Known bleeding diathesis or coagulation disorder
10. Presence of intracardiac lead in the right ventricle or right atrium
11. Presence of intracardiac thrombus
12. Major trauma within the past 14 days
13. Cardiovascular or pulmonary surgery within last 7 days
14. Known serious, uncontrolled sensitivity to radiographic agents
15. Contraindication to anticoagulants, i.e., heparin or alternative
16. Patient on extracorporeal membrane oxygenation (ECMO)
17. Cancer requiring active chemotherapy
18. Heparin-induced thrombocytopenia (HIT)
19. Pulmonary hypertension with peak pulmonary artery pressure >70 mmHg by right heart catheterization.
20. History of chronic severe pulmonary hypertension, and/or chronic left heart disease with left ventricular ejection fraction ≤30%
21. Life expectancy <90 days as determined by investigator
22. Pregnant or nursing
23. COVID-19 positive at hospital admission
24. Current participation in another investigational study
25. Evidence such as imaging or other that suggests the subject is not appropriate for this procedure (e.g., target vessel size is too small to accommodate 16F or 24F catheters).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Rate of major adverse events | 48 hours
  Major bleeding, device-related mortality, device-related serious adverse events
Mean reduction of RV/LV ratio | Baseline to 48 hours
  Change in RV/LV ratio from baseline to post procedure assessed by CT Angiography and adjudicated by an independent Core-lab

SECONDARY OUTCOMES:
Rates of Major bleeding, device-related mortality, device-related clinical deterioration, device-related pulmonary vascular injury and device-related cardiac injury | 48 Hours
  Evaluate rates of major bleeding, device-related mortality, device-related clinical deterioration, device-related pulmonary vascular injury and device-related cardiac injury
Rates of PE related mortality, all-cause mortality, device-related SAEs and symptomatic PE recurrence | 30 Days
  Evaluate rates of PE related mortality, All-cause mortality, Device-related SAEs and Symptomatic PE recurrence

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Huntsville Hospital, Huntsville, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Endeavor Health, Glenview, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ascension St John Hospital, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Northwell Health, Mount Kisco, New York
  - NYU Grossman School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Bon Secours Mercy Health, Inc, Cincinnati, Ohio
  - Prisma Health, Greenville, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - Medical City Fort Worth Hospital, Fort Worth, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

REFERENCES:
- [Derived] Bangalore S, Tomalty RD, Kado H, Sayfo S, Raskin A, Qamar A, Vargas Estrada A, Garcia-Reyes K, Lipshutz HG, Yallapragada S, Butty S, Gandhi S, Dexter D, Trivax J, Ali F, Knox M, Ramos C, Al-Saghir Y, Bishay V. Prospective Multicenter IDE Study of the Next-Generation Precision Aspiration Thrombectomy System for Intermediate-Risk Pulmonary Embolism: The SYMPHONY-PE Trial. Circ Cardiovasc Interv. 2025 Nov;18(11):e015815. doi: 10.1161/CIRCINTERVENTIONS.125.015815. Epub 2025 Sep 17. PMID 40961960